CLINICAL TRIAL: NCT00897273
Title: Human Papillomavirus Infection of the Mouth in Young Men and Risk Factors for Oropharyngeal Cancer
Brief Title: Oral HPV Infection in Young Men
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J0729; P30CA006973 (NIH); NA_00009472 (Other: JHM IRB); JHOC-J0729; CDR0000554422 (Other: other)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2013-04

CONDITIONS: Head and Neck Cancer; Infection; Precancerous Condition
Keywords: recurrent squamous cell carcinoma of the oropharynx; oropharyngeal cancer; oropharyngeal squamous cell carcinoma; infection; precancerous condition; human papilloma virus infection
MeSH Terms: conditions — Head and Neck Neoplasms; Infections; Precancerous Conditions; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Papillomavirus Infections | interventions — Comparative Genomic Hybridization; Gene Expression Profiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory Methods:
  Oral rinse sample:
  Standard, well-validated assays will be used to detect HPV genomic DNA in oral exfoliated cells from the Scope oral rinse sample.
  Serum sample:
  Standard laboratory assays will be used to detect antibodies to HPV16 L1 viral capsid protein.

INTERVENTIONS:
Genetic: comparative genomic hybridization
Genetic: gene expression analysis
Other: study of socioeconomic and demographic variables
Procedure: evaluation of cancer risk factors
Procedure: study of high risk factors

SUMMARY:
RATIONALE: Gathering information about human papillomavirus infection of the mouth in young men may help doctors learn more about risk factors for oropharyngeal cancer.

PURPOSE: This research study is assessing human papillomavirus infection of the mouth in young men and risk factors for oropharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the prevalence of oral human papillomavirus (HPV) type 16, 18, 6, or 11 infection in young adult men.
* Assess the independent effect of distinct sexual practices, including kissing, oral sex, and vaginal intercourse, on oral HPV prevalence.
* Estimate the 6-month incidence of HPV infection in this study population.

OUTLINE: Participants are assessed for oral human papillomavirus virus (HPV) infection (i.e., types 16, 18, 6, and 11) and for known or potential risk factors associated with the infection, including sexual behavior (e.g., kissing, performing oral sex, or vaginal intercourse), demographic characteristics (e.g., age or race), and history of HPV or other sexually transmitted infections. Prior exposure to HPV vaccine is also assessed.

Oral rinse samples are collected from participants at baseline and at 6 months for detection of HPV genomic DNA in oral exfoliated cells. Baseline serum samples are also collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently enrolled at one of the following institutions:

  * Johns Hopkins University
  * University of Maryland
  * Towson University

PATIENT CHARACTERISTICS:

* Able to understand the procedures and the potential risks involved as determined by clinic staff

PRIOR CONCURRENT THERAPY:

* No prior Gardasil® off label

Ages: 18 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience sample of 500 men recruited from Baltimore-area college health centers (Johns Hopkins University, University of Maryland, or Towson University).
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05-05 (Actual)

PRIMARY OUTCOMES:
Presence of an oral human papillomavirus (HPV) type 16, 18, 6 or 11 infection | 2 years
Presence of oral HPV infection by any of 37 HPV types | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maura Gillison, MD, PhD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins

REFERENCES:
- [Result] Gillison ML. Human papillomavirus-related diseases: oropharynx cancers and potential implications for adolescent HPV vaccination. J Adolesc Health. 2008 Oct;43(4 Suppl):S52-60. doi: 10.1016/j.jadohealth.2008.07.002. PMID 18809146
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials